CLINICAL TRIAL: NCT03874819
Title: Effect of an eXtended Permeability DiAlysis MembraNe on ESA Resistance in HemoDialysis Patients
Brief Title: Effect of a Medium Cut-Off Dialyzer - Medical Device on ESA Resistance in 110 Hemodialysis Patients (EXPAND)
Acronym: EXPAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carlo Maria Guastoni (Other)
Responsible Party: Sponsor-Investigator, Carlo Maria Guastoni, Head of Operative Unit of Dialysis and Nephrology, Azienda Ospedaliera, Ospedale Civile di Legnano
Organization: Azienda Ospedaliera, Ospedale Civile di Legnano (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EXPAND
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional Hemodialysis using a high-flux dialyzer
  Interventions: Device: High-flux dialyzer
- Experimental group (Experimental): Conventional Hemodialysis using a medium cut-of dialyzer
  Interventions: Device: Medium cut-off dialyzer

INTERVENTIONS:
Device: Medium cut-off dialyzer — Treatment using a Medium Cut-Off Dialyzer
  Arms: Experimental group
Device: High-flux dialyzer — Treatment using a high-flux dialyzer
  Arms: Control group

SUMMARY:
It is hypothesized that a consistent use of Medium cut-off membrane (Theranova) increased clearance of pro-inflammatory molecules in a broad molecular weight range attenuates the chronic inflammatory state in patients with poor response to ESA therapy and absence of absolute iron deficiency and that this leads to an improvement in ESA responsiveness (EPO resistance index).

DETAILED DESCRIPTION:
Hemodialysis Patients present chronic inflammation caused by multiple inflammatory stimuli. Chronic inflammation is linked to clinical signs and symptoms and cardiovascular mortality in these patients. Inflamed dialysis patients show impaired response to erythropoiesis-stimulating agents (ESA) mainly related to a reduced iron utilization (functional iron deficiency) with a greater need for ESA to meet hemoglobin targets. If absolute iron deficiency can been excluded, EPO resistance is likely related to 'inflammatory block'.

The high molecular permeability of the Theranova Medium cut-off membrane allows for significant clearance of medium molecular toxins and we know that a number of uremic solutes have been identified as pro-inflammatory, including several with a molecular weight in the size range of 20-45 kDa (cytokines, kappa/lambda free light chains and hepcidine). The EPO index has been previously used in clinical trials to measure EPO responsiveness [2,3] and is associated with mortality of ESRD patients [4-7].

All AE, SAE and other safety issues will be collected and described. The even review committee could be consulted in case of Safety event, and give recommendations.

Data entry to be carried out into an electronic CRF hosted database. This database allows the follow-up of any modifications made during data entry and monitoring. Data consistency will be checked on line according to the procedure described in the Data Management Plan (DMP), as part of the Study Master File. Each eCRF follows the study schedule structure. It is divided in sections for each visits or specific forms.

Eligible patients will be consecutively randomized in a 1:1 fashion to the standard dialysis or to dialysis with MCO dialyzer. The random sequence will be centrally generated in the CRF tool. The randomization procedure will be stratified per centre. Size of block is only known by the statistician to keep the investigator blinded regarding group allocation for the next patient.

Each patient must be identified on the CRF with his initials and identification number. Investigators must keep the list of all the patients, including identification numbers, full names and last known addresses.

Patients must be informed that the results obtained will be computer-stored and analyzed, that local laws must be applied, that patient's confidentiality must be preserved, and that they are entitled to obtain any information concerning the data stored and analyzed by a computerized system.

The investigator must give the Study Monitor direct access to relevant hospital or clinical records to confirm their consistency with the CRF entries. No information in these records about the identity of the subjects will leave the study site. Standards requirement is full verification for the presence of informed consent, adherence to the inclusion/exclusion criteria, documentation of SAEs and the recording of primary efficacy and safety variables. Additional checks of the consistency of the source data with the CRFs are performed according to the study-specific monitoring plan.

The final statistical analysis will be described in the Statistical Analysis Plan (SAP), which will be prepared and signed prior to clean file. The SAP will include detailed information regarding the analysis of safety and efficacy. Per protocol dataset will be defined by Endpoint Review Board.

Considering these assumptions, it is estimated that 55 patients per group will be required for a mean follow- up period of 48 weeks. A total number of 110 patients is required.

Continuous variables will be analyzed by ANOVA for repeated measurements. Data will be expressed as mean standard deviation if normally distributed or as percentile of the distribution elsewhere for continuous variables and as proportion for dichotomous variables.

The investigators must keep essential study documents (including all original raw data together with the patients' identification list and signed informed consents) minimum 5 years after product commercialization is stopped and should be retained for a longer period however if required by the applicable regulatory requirements or by an agreement with the sponsor.

Patient medical files have to be kept as much as possible at each investigation site.

Investigators will be informed by Sponsor when documents related to the study could be deleted. Prior to destroying study-related documentation, the investigator shall make sure with the Sponsor, which it does not need to be kept any longer.

Results of this clinical study will be submitted to a respected international peer-reviewed journal. They may also be submitted as abstracts to a scientific congress for oral or poster communication.

ELIGIBILITY:
Inclusion Criteria:

1. ESRD treated with chronic HD for at least 3 months
2. Treatment with high flux dialyzers for at least 3 months
3. Age ≥18 years
4. Receiving intravenous short acting ESA to treat anemia for at least 3 months
5. Impaired ESA responsiveness as indicated by EPO resistance index >median of patients in study center
6. transferrin saturation (TSAT) ≥20% (last routine value prior to randomization)
7. serum ferritin ≥100 ng/ml (last routine value prior to randomization)
8. Signed informed consent.

Exclusion Criteria:

1. Acute infection ≤4 weeks prior to randomization
2. HIV or hepatitis infection
3. Central Venous Catheter (with the history of infections in the latest 3 months)
4. chronic liver disease
5. active cancer
6. known blood dyscrasia (paraprotein abnormalities)
7. known bleeding disorders
8. Bleeding episode ≤12 weeks prior to randomization
9. Blood/red cell transfusion ≤12 weeks prior to randomization
10. hypoalbuminemia defined as serum albumin concentration below 35 g/L
11. (last routine value prior to randomization)
12. Participation in another clinical interventional investigation
13. Pregnancy
14. Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Change of the "Erythropoietin Responsiveness factor" (EPO index) | Up to 48 weeks
  EPO index will be calculated as the average weekly EPO dose in IU per kg BW in the preceding 4 weeks divided by the last measured Hb

SECONDARY OUTCOMES:
Inflammation status | Up to 48 weeks
  Evaluation of predialysis plasma values every 8 weeks of: FLCs (kappa and lambda), CRP, Hepcidin.
Metabolic diseases | Up to 48 weeks
  Evaluation of predialysis plasma values every 8 weeks of: urea, beta 2 microglobulin, myoglobin and albumin